CLINICAL TRIAL: NCT00417560
Title: A Single Center, Open-label, Phase I/II Study of Two 90 Microgram Doses of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Adult Subjects at Risk of Occupational Exposure to Live H5N1 Viruses
Brief Title: Inactivated Influenza A/H5N1 Vaccine in Adult Subjects at Risk of Occupational Exposure to Live H5N1 Viruses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDC-NCIRD-5000
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Influenza
Keywords: Influenza A/H5N1 vaccine avian influenza H5N1 H5N1
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Experimental: Influenza A/H5N1 Vaccine (Experimental): Two 90ug Doses of Intramuscular Inactivated Influenza A/H5N1 Vaccine
  Interventions: Biological: inactivated influenza A/H5N1 vaccine

INTERVENTIONS:
Biological: inactivated influenza A/H5N1 vaccine

SUMMARY:
This is a single center, open-label, Phase I/II study in up to 100 adult subjects, aged 18 years and older who are at occupational risk of exposure to live H5N1 viruses. This study is designed to investigate the safety, reactogenicity, and immunogenicity of two 90 µg doses of an investigational inactivated influenza A/H5N1 virus vaccine given approximately 28 days apart. A blood sample will be collected for immunogenicity evaluation prior to each vaccination. Subjects will maintain a memory aid (appendix C4 and C13) to record oral temperature and systemic and local AEs for 7 days after immunization. Subjects will be encouraged to take their temperature around the same time each day. All subjects will receive a safety follow-up telephone call at 1 to 3 days after each vaccination (approximately Day 2) to elicit any AE and concomitant medication information. Subjects will return to the clinic 7 days after each vaccination for assessment of AEs and concomitant medications, a targeted physical examination (if indicated), and review of the memory aid. At approximately Day 28 after the first vaccination, subjects will return to the clinic for evaluation of vital signs, blood sample collection and safety follow-up, confirmation of eligibility criteria and a second vaccination. Safety follow-up will be identical to that performed after the first vaccination. At approximately Day 56 (or about 28 days after the second vaccination), subjects will return to the clinic for immunogenicity blood sample collection, AE and concomitant medication assessment, and targeted physical examination and vital sign assessment (if indicated). At approximately Day 180 (6 months after the first vaccination), subjects will return to the clinic for a final immunogenicity blood sample collection and safety assessment.

DETAILED DESCRIPTION:
* This is a single center, open-label, Phase I/II study in up to 100 adult subjects, aged 18 years and older who are at occupational risk of exposure to live H5N1 viruses. This study is designed to investigate the safety, reactogenicity, and immunogenicity of two 90 µg doses of an investigational inactivated influenza A/H5N1 virus vaccine given approximately 28 days apart. A blood sample will be collected for immunogenicity evaluation prior to each vaccination. Subjects will maintain a memory aid (appendix C4 and C13) to record oral temperature and systemic and local AEs for 7 days after immunization. Subjects will be encouraged to take their temperature around the same time each day. All subjects will receive a safety follow-up telephone call at 1 to 3 days after each vaccination (approximately Day 2) to elicit any AE and concomitant medication information. Subjects will return to the clinic 7 days after each vaccination for assessment of AEs and concomitant medications, a targeted physical - Page 2 of 5 - examination (if indicated), and review of the memory aid. At approximately Day 28 after the first vaccination, subjects will return to the clinic for evaluation of vital signs, blood sample collection and safety follow-up, confirmation of eligibility criteria and a second vaccination. Safety follow-up will be identical to that performed after the first vaccination. At approximately Day 56 (or about 28 days after the second vaccination), subjects will return to the clinic for immunogenicity blood sample collection, AE and concomitant medication assessment, and targeted physical examination and vital sign assessment (if indicated). At approximately Day 180 (6 months after the first vaccination), subjects will return to the clinic for a final immunogenicity blood sample collection and safety assessment. Blood samples collected prior to each vaccination (Days 0 and 28) and on Days 56 and 180 after the first vaccination will be tested at the CDC Influenza Division Laboratory for the levels of neutralizing and HAI antibodies and CMI responses. The primary outcome measures will be the frequencies and severities of AEs and the GMTS and proportions of subjects who achieve 4-fold rises in serum neutralizing and HAI titers against the influenza A/H5N1 virus on Day 56. Serum HAI and neutralizing antibody responses (including frequencies of 4 fold or greater rise in titer; GMTs; and proportions of subjects achieving protective titers of neutralizing antibody 1 month and 6 months after first dose) will also be assessed. A secondary outcome measure will be CMI responses evaluated 1 month after the receipt of each dose of vaccine and 6 months after the receipt of the first dose of vaccine

ELIGIBILITY:
Inclusion Criteria

* Non-pregnant
* Non-immune compromised adults 18 years and older
* At occupational risk of exposure to live H5N1 viruses
* Must be eligible for care by the CDC occupational health clinic

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bridges, MD, Principal Investigator — Centers for Disease Control and Prevention